CLINICAL TRIAL: NCT04669184
Title: Assessment of Sarcopenia, Physical Performance and Cognitive Function in Hemodialysis Patients
Brief Title: Sarcopenia and Physical Performance in Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Firat, Principal Investigator, Hacettepe University
Other Study IDs: GO 20/338
Record Dates: First submitted 2020-07-03; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: End Stage Kidney Disease
Keywords: sarcopenia; pain; physical performance
MeSH Terms: conditions — Kidney Failure, Chronic; Sarcopenia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Many systems such as the cardiovascular, pulmonary, musculoskeletal, hematological, immunological, gastrointestinal, central nervous system are affected due to decreased kidney function. The aim of this study was to investigate the relationship between physical performance and sarcopenia, peripheral muscle strength, activities of daily living, cognitive functions, physical activity level, fragility, pain in hemodialysis patients.

DETAILED DESCRIPTION:
A high prevalence of sarcopenia has been reported in end stage kidney disease. The incidence of sarcopenia increases with age. Muscle atrophy is caused by an imbalance between the anabolic and catabolic processes in chronic kidney disease. Sarcopenia and physical inactivity progress synergistically. Decreased physical performance is associated with sarcopenia. In hemodialysis patients, daily physical activity level and physical performance decrease. Cognitive impairment is common in chronic kidney disease. Uremic toxins can cause a decrease in cognitive function. One of the most important problems associated with hemodialysis is pain and pain negatively affects functional capacity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with end stage kidney disease
* Receiving hemodialysis for more than 3 months
* Being clinically stable
* Volunteering to participate in the research

Exclusion Criteria:

* Having an orthopedic disease that may affect functional capacity
* Having cardiac event in the past 3 months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older, who are diagnosed with end stage kidney disease at the Hacettepe University, Faculty of Medicine, Department of Internal Diseases, Nephrology Subdivision
Sampling Method: Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Sarcopenia | 5 minutes
  Sarcopenia will be evaluated using SARC-F questionnaire. For SARC-F, a total score of ≥ 4 indicates sarcopenia.
Physical performance will be evaluated using Short physical performance battery. | 10 minutes
  The total score of Short physical performance battery ranges from 0 to 12.
Physical performance will be evaluated using 1 minute sit to stand test. | 5 minutes
  1 minute sit to stand test, the maximum number of repetitions within the established time was recorded
Pain level | 5 minutes
  Pain will be evaluated using Short-form McGill Pain questionnaire

SECONDARY OUTCOMES:
Peripheral muscle strength | 5 minutes
  Knee extensor and hand grip strength will be evaluated using dynamometer.
Cognitive function | 10 minutes
  Cognitive function will be evaluated using Standardized Mini-Mental State Examination. The test is a 30-point screening tool. Higher scores mean a better outcome.
Physical activity level | 5 minutes
  Physical activity level will be evaluated using International Physical Activity Questionnaire-Short Form
Fragility | 5 minutes
  Fragility will be evaluated using the five Fried frailty criteria (unintentional weight loss, exhaustion, weakness, slowness, low physical activity). The total score is interpreted as follows: 0 non-frail, 1-2 pre-frail and 3-5 frail
Activities of daily living | 10 minutes
  Activities of daily living will be evaluated using Barthel Index for Activities of Daily Living.The total score is100 and higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Firat, MSc, Principal Investigator — Hacettepe University; Naciye Vardar-Yagli, PhD, Study Director — Hacettepe University; Deniz İnal-İnce, Professor, Study Chair — Hacettepe University; Tolga Yildirim, MD, Study Chair — Hacettepe University; Melda Saglam, PhD, Study Chair — Hacettepe University; Ebru Calik-Kütükcü, PhD, Study Chair — Hacettepe University